CLINICAL TRIAL: NCT03518229
Title: Pilot Study of Intervention to Reduce Sunburns in Melanoma Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Converted from a pilot into a larger study which we will enter as a new protocol
Sponsor: University of Minnesota (Other)
Collaborators: Melanoma Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00002107
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Melanoma (Skin)
Keywords: cancer prevention; sunburn
MeSH Terms: conditions — Melanoma; Sunburn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Microsoft Band 2 application with UV messaging activated
  Interventions: Device: Microsoft Band 2 + UV messaging
- Control (Active Comparator): Microsoft Band 2 application (UV messaging not active)
  Interventions: Device: Microsoft Band 2

INTERVENTIONS:
Device: Microsoft Band 2 + UV messaging — wearable device (wrist) and associated mobile application; UV sensor and messaging activated
  Arms: Intervention
Device: Microsoft Band 2 — wearable device (wrist) and associated mobile application; UV messaging not activated
  Arms: Control

SUMMARY:
This project will pilot test whether a wearable device that tracks sun exposure and provides alerts regarding sun exposure and protection behaviors will reduce sunburns in melanoma survivors. The use of wearable technology devices has grown quickly over the last decade and studies using these devices to promote physical activity and weight loss have been promising. The investigators will pilot test the technology device versus a similar control device in 80 melanoma survivors and compare sunburns between the two groups after the three month intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Diagnosed with stage I-III cutaneous invasive melanoma between 2009 and 2017 and treated at the University of Minnesota
* Able to read/write in English
* Own a smartphone
* Able to provide voluntary informed consent

Exclusion Criteria:

-Patients currently undergoing adjuvant therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Sunburn | 3 months
  Self-report of a sunburn during study period

IPD SHARING:
Plan to Share IPD: No